CLINICAL TRIAL: NCT04458532
Title: A Randomized Trial to Minimize Non-Response to Aerobic Training in Post-Menopausal Women With Early Stage Breast Cancer
Brief Title: Exercise Therapy to Improve Cardiovascular Health in Post-Menopausal Women After Treatment for Early Stage Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-130
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Early Stage Breast Cancer
Keywords: Exercise Therapy; Aerobic Training; Post-Menopausal Women; 20-130

STUDY DESIGN:
Intervention Model Description: This is a single-center randomized controlled trial (RCT) study designed to evaluate the cardiorespiratory fitness (CRF) response rate to different aerobic therapy (AT) doses in patients with post-treatment primary breast cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- (A) breast cancer after completion of chemo (Experimental): 300 min/wk for 16 weeks, followed by 16 weeks of usual care.
  Interventions: Other: Aerobic Training
- (B) breast cancer after completion of chemo (Experimental): 150 min/wk for 32 weeks.
  Interventions: Other: Aerobic Training
- (C) breast cancer after completion of chemo (Experimental): 300 min/wk for 32 weeks.
  Interventions: Other: Aerobic Training
- (D) breast cancer after completion of chemo (Active Comparator): 150 min/wk for 16 weeks, followed by 16 weeks of usual care.
  Interventions: Other: Aerobic Training

INTERVENTIONS:
Other: Aerobic Training — 300 min/wk for 16 weeks
  Arms: (A) breast cancer after completion of chemo
Other: Aerobic Training — 150 min/wk for 32 weeks
  Arms: (B) breast cancer after completion of chemo
Other: Aerobic Training — 300 min/wk for 32 weeks
  Arms: (C) breast cancer after completion of chemo
Other: Aerobic Training — 150 min/wk for 16 weeks
  Arms: (D) breast cancer after completion of chemo

SUMMARY:
This study will compare the effects on cardiorespiratory fitness (CRF) of aerobic exercise in different amounts (number of minutes/session) over different periods of time (number of weeks). Aerobic exercise is physical activity of light-to-moderate intensity that uses the large muscle groups (muscles in your legs, buttocks, back, and chest) and can be performed for at least 10 minutes.

The researchers will study the effects of different exercise programs on how well the study participants' bodies use oxygen, how well their heart pumps blood, how well their lungs function, and how healthy their blood vessels are.

DETAILED DESCRIPTION:
Prior to the initiation of every supervised aerobic training session, patient resting vital signs will be assessed to ensure the patient can safely proceed with the session. Vital signs, including resting heart rate and blood pressure, will be collected and monitored per ExOnc program guidelines. In addition, the planned session will not be initiated if the ExOnc staff member observes any concerns that may compromise participant safety and/or the integrity of the planned session. Vital sign monitoring guidelines for unsupervised sessions, prescribed at lower intensities, will be advised by the exercise physiologist at the time the session plan is provided to the patient. Patients will be instructed to not begin an unsupervised session if their resting heart rate or blood pressure is outside the recommended guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-80 years
* Female
* Surgically resected early stage (I-III) primary breast cancer
* Post-menopausal, defined as one of the following:

  * Age ≥ 45 with no menses for at least 2 years
  * Chemically and/or surgically induced menopause through ovarian suppression, as determined by the primary oncologist
  * Estradiol level of ≤30 pg/mL
* An interval of at least one year, but no more than five years, following the full completion of definitive therapy for malignant disease. Definitive therapy is defined as:

  * Surgery plus radiation
  * Surgery plus chemotherapy
  * Surgery plus trastuzumab
* Exercise intolerance (i.e., patients must have a VO2peak below the predicted for active age and sex-matched individuals. (+/- the technical error of 1.32 mL/kg/min)].

Note: Normative values are available up to 80 years of age)

* Able to complete an acceptable baseline CPET, in the absence of high-risk ECG findings or other inappropriate response to exercise as determined by the PI, as defined by any of the following criteria:

  * Achieving a plateau in oxygen consumption, concurrent with an increase in power output;
  * A respiratory exchange ratio ≥ 1.10;
  * Attainment of maximal predicted heart rate (HRmax) (i.e., within 10 bpm of age-predicted HRmax [HRmax = 220-Age[years]);
  * Volitional exhaustion, as measured by a rating of perceived exertion (RPE) ≥ 18 on the BORG scale
* Willingness to comply with all study-related procedures.

Exclusion Criteria:

* Any of the following absolute contraindications to cardiopulmonary exercise testing:

  * Acute myocardial infarction within 3-5 days of any planned study procedures
  * Unstable angina
  * Uncontrolled arrhythmia causing symptoms or hemodynamic compromise
  * Recurrent syncope
  * Active endocarditis
  * Acute myocarditis or pericarditis
  * Symptomatic severe aortic stenosis
  * Uncontrolled heart failure
  * Acute pulmonary embolus or pulmonary infarction within 3 months of any planned study procedures
  * Thrombosis of lower extremities
  * Suspected dissecting aneurysm
  * Uncontrolled asthma
  * Pulmonary edema
  * Respiratory failure
  * Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (e.g., infection, renal failure, thyrotoxicosis)
* Presence of any other concurrent, actively treated malignancy
* History of any other malignancy treated within the past 3 years (other than non-melanoma skin cancer)
* Presence of distant metastatic disease (i.e., stage IV)
* Room air desaturation at rest ≤ 85%
* Mental impairment leading to inability to cooperate.
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the participant a poor candidate for the trial.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Post-Menopausal Women After Treatment for Early Stage Breast Cancer
Enrollment: 152 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
peak oxygen consumption (VO2peak; ml O2.kg-1.min) response rate | 32 weeks
  A CRF change ≥1.32 ml O2.kg-1.min-1 will be considered a response; a change <1.32 ml O2.kg-1.min-1 will be considered a non-response.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital (Data Collection Only), Hartford, Connecticut
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm